CLINICAL TRIAL: NCT05711004
Title: Efficacy of Education Via Phone-based Text Messaging (SMS) on Patients With Uncontrolled Hypertension: a Randomized Controlled Trial
Brief Title: Efficacy of Education Via Phone-based Text Messaging (SMS) on Patients With Uncontrolled Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Reza Safarpour, Manager in chief of gastroenterohepatology research center, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 27586
Record Dates: First submitted 2023-01-14; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Eligible participants with uncontrolled HTN will be randomly assigned to experiment (SMS) or control (routine care) groups at a 1:1 ratio.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS group (Experimental): Participants in the experimental group will receive three messages per week in the morning (9-10 am) for three months. The investigators will call them every month to ensure that the SMS is delivered.
  Interventions: Behavioral: Education via SMS
- Control group (No Intervention): Patients in the control group will also receive the usual primary health care.

INTERVENTIONS:
Behavioral: Education via SMS — Participants in the experimental group will receive three messages per week in the morning (9-10 am) for three months. The investigators will call them every month to ensure that the SMS is delivered.
  Arms: SMS group

SUMMARY:
Uncontrolled hypertension (HTN) is a major public health worldwide, which increases the risk of cardiovascular diseases. Low adherence to medication, unhealthy lifestyle and poor knowledge of HTN diagnosis and treatment are among the known factors associated with uncontrolled HTN. Digital innovations became popular as low-cost tools to provide personalized advice to people with long-term health conditions, leading to their adherence to health behavior modifications. Therefore, this randomized single-blind controlled trial (RCT) aimed to test whether providing health information via a short message service (SMS) influences blood pressure control, health practice, and medication adherence. For the current RCT, the investigators will use data from the PERSIAN Kavar cohort study (PKCS). Eligible participants with uncontrolled HTN will be randomly assigned to experiment (SMS) or control (routine care) groups at a 1:1 ratio. Participants in the experimental group will receive three messages/per week for three months. Systolic and diastolic blood pressure will be the primary outcomes of this study. Medication adherence and practice related to cardiovascular diseases will the secondary outcomes. These variables will be assessed before and after the intervention. At the end of the study, the acceptability of the messages will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a diagnosis of HTN by a clinician at the baseline or until the third follow-up of PKCS, have uncontrolled HTN (≥140/90) at the enrollment, have a prescription for blood pressure-lowering medication, understand Persian, have regular access to a mobile phone, and are able to read SMS by themselves or with their family's help. The investigators will enroll only one member per household.

Exclusion Criteria:

* Those with renal failure or requiring specialist care for their hypertension at a hospital, pregnant women or who are within 3 months postpartum, patients with severe physical or mental illness, and subjects not willing to participate in the study.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Three months after the start of intervention
  Systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Medication adherence which will be assessed by Morisky Medication Adherence Scale | Three months after the start of intervention
  Adherence to the anti-HTN drugs will be assessed by Morisky Medication Adherence Scale .
Practice according to the KAP questionnaire | Three months after the start of intervention
  The questions of "Knowledge, Attitude, and Practice Regarding Cardiovascular Diseases" (doi: 10.5812/ijem.101612) questionnaire that are related to Practice will be completed for patients.
Weight | Three months after the start of intervention
  Body weight (kg)
Number of patients who think that messages were usefull and had positive impact | Three months after the start of intervention
  Acceptability of the messages will be assessed according to the questiones listed in doi: 10.5334/gh.1103

IPD SHARING:
Plan to Share IPD: Undecided